CLINICAL TRIAL: NCT05558020
Title: Feasibility of Constant Work Rate Testing to Detect Exercise-induced Laryngeal Obstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Emil Walsted, Principal Investigator, Bispebjerg Hospital
Other Study IDs: H-20057391
Record Dates: First submitted 2022-09-15; First posted 2022-09-28 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Exercise-induced Laryngeal Obstruction (EILO)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Continuous laryngoscopy during exercise (CLE), incremental exercise protocol — The incremental work rate exercise test will be performed using a cycle-ergometer. The exercise protocol is initiated by a five-minute warm-up at 50 Watts (W). Subsequently, they will complete a stepwise protocol, which will begin at 100 W and increase by 2 W every 6th second, until exhaustion or until the patient is unable to continue exercise, for any reason.
Diagnostic Test: Continuous laryngoscopy during exercise (CLE), continuous work rate protocol — Within two weeks the participants will perform an additional CLE-test at various intensities. The new exercise protocol is designed to induce EILO at different exercise intensities. Using the participants' individually calculated exercise capacity, three different workloads (70 %, 80 % and 90 %) will be calculated.
  The exercise protocol will be initiated with a five-minute warm-up at 50 W, then the workload will increase to the watt equivalent to 70 % of the participant's maximal exercise capacity. This workload will be fixed for ten minutes and only terminated if the participant feels the need to stop due to exhaustion or breathing difficulties. Next, the participant will have a five-minute resting phase with a set workload of 50 W. This protocol will be repeated at a workload equivalent to 80 % and 90 %

SUMMARY:
TITLE Feasibility of constant work rate testing to detect exercise-induced laryngeal obstruction

DESIGN Prospective observational pilot study

AIMS To investigate if constant work rate testing at different work rates will sufficiently induce detectable exercise-induced laryngeal obstruction (EILO) using CLE.

POPULATION Adult patients with EILO

DURATION 01.09.2022 - 30.06.2023

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 or above with a clinical suspicion of having EILO.
* Individuals with concurrent asthma can participate in the study provided that their asthma is well-controlled, determined by a negative bronchoprovocation test.

Exclusion Criteria:

* No EILO found in Clinical standard-of-care CLE test
* Not able to complete the exercise test for other reasons than breathlessness or leg fatigue (e.g. injury, disease or disability preventing cycling to maximal exertion).
* Comorbidities other than asthma, which, judged by the investigator, might confound the test results or pose a medical risk to the patient (e.g. cardiac disease, exercise-induced anaphylaxis).
* Current smokers (< 6 months of stopping) or individuals with a significant smoking history (>10 pack years).
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals referred to CLE testing at the asthma service at Bispebjerg Hospital in Copenhagen, Denmark, for the investigation of exercise-related respiratory symptoms, will be offered to participate in the present study in addition to the standard-of-care incremental CLE test.
  Al patients will be evaluated during the visit to the asthma service at Bispebjerg Hospital to ensure they are clinically fit for exercise testing.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
prevalence and degree of glottic or supraglottic collapse in EILO patients | Changes from baseline during the procedure and immediately after cessation of the exercise test.
  Laryngoscopic detection of supraglottic or a glottic obstruction of the same severity as observed during incremental testing, during a submaximal constant work rate exercise test (70 %, 80 % and 90 %) using a visual grade scale (0-3, with 0 reflecting no obstruction, and 3 being the most severe degree of obstruction).
Time of onset of the laryngeal obstruction | A time of onset determined during the procedures
  A specific point in time where observed laryngeal obstruction is first discernible will be determined during the evaluation of the laryngoscopic videos.
  This is to descriptively quantify this outcome.
Observed duration of the laryngeal obstruction | Duration measured in seconds during the procedures
  The investigators will further evaluate the laryngoscopic videos and determine the duration of the participant's laryngeal obstruction. This duration is defined as the time period from the time of onset during submaximal exercise, until remission of the observed obstruction or end of the test.

SECONDARY OUTCOMES:
Patient reported symptom score: Dyspnoea-12 | At baseline
  The patients will fill out the Dyspnoea-12 questionnaire before the first exercise test The questionnaire consists of 12 questions regarding dyspnoea. This is a descriptive measure
Patient reported symptom scores: Nijmegen | At baseline
  The participants will fill out the Nijmegen questionnaire before the first exercise test The questionnaire consists of 16 questions, with answers ranging from "never" to "very often". A score is calculated from these answers. A higher score means that it is more likely that the participant suffers from hyperventilation syndrome.
  This is a descriptive measure
Patient reported symptom scores: Multidimensional Dyspnoea Profile (MDP). | At baseline
  The patients will fill out the Multidimensional Dyspnoea Profile (MDP) questionnaire before the first exercise test This profile consists of questions regarding both affective and sensory components of dyspnoea.
  This is a descriptive measure
Modified borg dyspnoea during exercise | At baseline and at one minute intervals during the CLE tests (up to 60 minutes)
  Minimum score: 0 Maximum score: 10 The participant will be asked to rate dyspnoea at baseline and during the CLE tests at 1 minute intervals.
  The investigators will compare the scores between the incremental CLE tests and the constant work rate CLE tests.
Leg fatigue scores during exercise | At baseline and at one minute intervals during the CLE tests (up to 60 minutes)
  Minimum score: 0 Maximum score: 10 The participant will be asked to rate leg fatigue at baseline and during the CLE tests at 1 minute intervals.
  The investigators will compare the scores between the incremental CLE tests and the constant work rate CLE tests.
Rate of perceived exertion (RPE) scores during exercise | At baseline and at one minute intervals during the CLE tests (up to 60 minutes)
  Minimum score: 0 Maximum score: 10 The participant will be asked to evaluate their rate of perceived exertion at baseline and during the CLE tests at 1 minute intervals.
  The investigators will compare the scores between the incremental CLE tests and the constant work rate CLE tests.
Inter-rater agreement of the prevalence and degree of glottic or supraglottic collapse in EILO patients | During data analysis (month 1).
  After obtaining laryngoscopic video data, the investigators will evaluate the severity of laryngeal obstruction using a visual grade scale (0-3).
  From these gradings we will calculate inter-rater agreement values (weighted kappa).

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, København NV, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thougaard J, Pedersen L, Walsted E. Feasibility of Constant Work Rate Testing to Detect Exercise-Induced Laryngeal Obstruction. Med Sci Sports Exerc. 2024 Mar 1;56(3):427-434. doi: 10.1249/MSS.0000000000003319. Epub 2023 Oct 12. PMID 38356163